CLINICAL TRIAL: NCT05755412
Title: Observational, Prospective, Single-arm Multicentric Study of Shockwave ®S4 Catheter IVL (Intravascular Lithotripsy) Balloon for the Treatment of Infrapopliteal Calcified Stenoses and/or Occlusions in Patients With Critical Limb Ischaemia
Brief Title: Shockwave ®S4 Catheter IVL to Treat Infrapopliteal Calcified Stenoses and/or Occlusions in CLTI Patients (LEGACY)
Acronym: LEGACY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EndoCore Lab s.r.l. (Other)
Collaborators: Fondazione Italiana Vascolare (Other)
Responsible Party: Sponsor
Other Study IDs: IVL012022
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease; Critical Limb-Threatening Ischaemia
Keywords: PAD; CLTI
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The study will evaluate the safety and efficacy of Peripheral Intravascular Lithotripsy system with Shockwave S4 catheter® for the treatment of de novo, re-stenosis or re-occlusive,calcified chronic total occlusion (CTOs) lesions in patients with Critical Limb Threatening Ischemia (CLTI).

DETAILED DESCRIPTION:
The present study is designed as a multicentre, prospective, single-arm, observational study.

All eligible subjects for undergoing intervention with Shockwave S4 catheter® Peripheral Intravascular Lithotripsy (IVL) at sites participating in the study will be considered for enrolment and will be asked to give consent prior to participating.

Subjects will be considered enrolled in the study at the time written informed consent is given to the use of their personal data. Once patients are enrolled, their demographics, medical history, disease-relevant conditions, treatment details and outcomes will be collected for up to 12 months from the procedure.

The study will collect information about the medical care patients receive during their planned procedure. No additional testing or procedures will be done.

The procedure with Shockwave S4 catheter® Peripheral Intravascular Lithotripsy (IVL) will be performed as per the current instructions for use.

After discharge all patients will attend clinic visits at 30 days (±14 days), 6 months (±30 days),12 months (±30 days).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient has signed an approved informed consent form
* Patient with Critical Limb Ischaemia, Rutherford category 4 (ischaemic rest pain), 5(minor tissue loss) or 6 (major tissue loss)
* Patient with Stenotic (>50% luminal loss) or occluded infrapopliteal artery, including the tibiofibular trunk, the anterior tibial artery, the posterior tibial artery and the peroneal artery
* The vascular lesion length will be no longer than 150 mm.
* Patient with no significant disease at the inflow: common iliac, external iliac, superficial femoral and popliteal artery on the ipsilateral side prior to enrollment, and patient with no significant disease at the outflow - runoff to ankle level: plantar for posterior tibial, pedal for anterior tibial, anterior and posterior perforant branches for peroneal vessels or previous successful revascularization of the disease segments (inflow-outflow)
* Live expectancy > 1 year.
* Presence at least ≥1 filling pedal vessel on the target limb.

Exclusion Criteria:

* Subject pregnant or planning to become pregnant during the study
* Subject no able to perform the follow up or other factors making clinical follow-up difficult
* Acute or Subacute limb ischaemia which requires thrombolysis as first treatment modality or previous thrombolytic therapy in the last 48-72 hours.
* Known allergy to concomitant medication, antiplatelet anti-coagulant or thrombolytic medication
* Poor inflow due to ipsilateral stenoses or occlusions of the iliac or femoropopliteal arteries
* Significant stenoses (> 50%) distal to the target lesion that might require revascularization or impede run-off
* Desert foot condition. No Patent foot main arteries
* Subject enrolled in another investigational study that has not reached its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by lower extremities artery disease and referred for the endovascular treatment of infrapopliteal calcified stenoses and/or occlusions in patients with critical limb ischaemia
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Composite of Acute Gain Index and freedom from clinically driven target lesion revascularization (CD-TLR) through 6 months post procedure | 30 days, 6 months
  Acute Gain Index defined as the Acute Gain (difference between the vessel diameter before and after IVL) divided by the Reference Vessel Diameter
  CD-TLR defined as as repeat percutaneous intervention or surgical bypass graft to treat an angiographic significant restenosis (>50%) at the level of the treated lesion ±10 mm (proximally and/or distally) in the presence of at least 1 of the following criteria:
  * recurrence of pain in the foot at rest that increases in the supine position
  * recurrence of pedal ulceration, evidence of halted healing
  * appearance of a new foot lesion
  * target vessel occlusion (by either angiography or DUS).

SECONDARY OUTCOMES:
Composite of Freedom from device and procedure-related death and freedom from target limb major amputation and clinically-driven and mechanical target lesion revascularization (CD-MTLR) | 30 days, 6 months
  Composite of Freedom from device and procedure-related death through 30 days post-procedure and freedom from target limb major amputation and clinically-driven and mechanical target lesion revascularization (CD-MTLR) through 6 months post-procedure
Late Lumen Loss Index | 6 months
  Late Lumen Loss defined as Late Lumen Loss divided by Acute Lumen Gain
Rutherford class shift | Baseline, 30 days, 6 months, 12 months
  Assess clinical improvement based on Rutherford class changes at 1, 6, 12 months, compared to baseline
Amputation rate | 30 days, 6 months, 12 months
  defined as rate of minor and major amputations
CD-TLR | 30 days, 6 months
  Clinically-driven target lesion revascularization (CD-TLR) is defined as any reintervention within the target lesion due to symptoms
Technical success | Day 1
  Technical success, defined as achievement of a final in-lesion residual diameter stenosis of ≤50% (as determined by the angiographic core lab), using the Shockwave S4 catheter, without a device malfunction after wire passage through the lesion.
Clinical Success | Day 1
  Clinical success (per subject) defined as technical success without the occurrence of major adverse events during the procedures (as determined by the angiographic core lab)
Procedural Success | Day 1
  Procedural success defined as lesion success without the occurrence of major adverse events during the procedure
Ankle-brachial index (ABI) or trans-cutaneous oximetry (TcPO2) improvements | Baseline,30 days, 6 months, 12 months
  Assess ABI or TcPO2 improvements
Major adverse event (MAE) rates | 30 days, 6 months, 12 months
  Major adverse event (MAE) rates, defined as the first occurrence of any of the following:
  death from any cause, major amputation (above-the-ankle) of the target limb and target lesion revascularization (TLR), through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariano L Palena, MD, Principal Investigator — Casa di Cura Abano Terme; Pierluigi Antignani, MD, Study Chair — Fondazione Vascolare Italiana; Gabriele Morselli, PharmD, Study Director — EndoCoreLab s.r.l.
Locations (4):
- Italy (4):
  - I.R.C.C.S. MultiMedica, Sesto San Giovanni, Milano
  - Casa di Cura Abano Terme, Abano Terme, Padova
  - Ospedale Pederzoli, Peschiera del Garda, Veneto
  - Arcispedale Santa Maria Nuova, Reggio Emilia